CLINICAL TRIAL: NCT03687034
Title: A Phase I Study of BRCX014 to Investigate Dose-Ranging Safety and Pharmacokinetics in Adults With Glioblastoma (GBM) and Non-Methylated MGMT Gene Status
Brief Title: A Study of the Safety and Pharmacokinetics of BRCX014 in Patients With Glioblastoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leaf Vertical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Olympian 2
Record Dates: First submitted 2018-08-22; First posted 2018-09-27 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: This study consists of dose escalations that follow the standard 3+3 design, proceeding until the maximum tolerated dose is attained. The treatment period for patients in this study at each dose will be one year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BRCX014 (Experimental): Subjects will receive escalating doses of BRCX014 in conjunction with standard-of-care (SOC) treatment. For patients with GBM, following standard chemo-radiation treatment (radiation: 2 Gy per day for a total of 60 Gy; and temozolomide: 75 mg per square meter of body-surface area per day, seven days per week from the first to the last day of radiotherapy), SOC treatment comprises six cycles of adjuvant temozolomide (150 to 200 mg per square meter for five days during each 28-day cycle), with or without use of alternating electric field therapy (Optune device).
  Interventions: Drug: Temozolomide; Device: Optune

INTERVENTIONS:
Drug: Temozolomide — Standard-of-care chemotherapy for patients with glioblastoma includes concurrent radiation therapy (2 Gy per day for a total of 60 Gy) and temozolomide (75 mg per square meter of body- surface area per day, seven days per week from the first to the last day of radiotherapy), followed by six cycles of adjuvant temozolomide (150 to 200 mg per square meter for five days during each 28-day cycle).
  Other Names: Temodar
Device: Optune — Standard-of-care treatment for glioblastoma includes alternating electric-field therapy, or Optune, as a Category 1 treatment in conjunction with temozolomide after maximal safe resection and completion of radiation therapy.
  Other Names: TTFields

SUMMARY:
An Open-Label, Multi-Center Study to Assess the Safety and Pharmacokinetics of BRCX014 Combined with Standard-of-Care Treatment in Subjects with Glioblastoma

DETAILED DESCRIPTION:
Several studies have shown a possible anti-tumor role for cannabinoids by modulating cell signaling pathways, inhibiting angiogenesis, inducing apoptosis, and overcoming chemotherapy resistance. The investigators seek to demonstrate the safety profile of BRCX014, a cannabinoid formulation, when given to glioblastoma patients in conjunction with standard-of-care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed glioblastoma (astrocytoma WHO grade IV)
* MGMT promoter methylation status is negative
* Brain MRI confirmation of disease according to RANO (Response Assessment in Neuro-Oncology) criteria
* Completion of standard-of-care temozolomide-based chemoradiation for post-operative treatment of glioblastoma plus two-to-six week "washout" period and stable-to-improved baseline brain MRI.
* Male and female subjects between the ages of 18 and 85 years
* Karnofsky Performance Score ≥ 60%
* Expected survival of at least six months from the day of enrollment
* No severe dysfunction of major organs (e.g., bone marrow, liver, kidneys, heart, lungs, etc.) and laboratory results from up to 14 days prior to enrollment fall within criteria:

  * Hemoglobin > 10 g/dL
  * Leukocytes ≥ 3,000 per μl
  * Absolute neutrophil count ≥ 1,500 per μl
  * Platelet count > 100,000 per μl
  * BUN < 25 mg
  * Serum creatinine within normal institutional limits OR Creatinine clearance ≥ 60 ml/min/1.73 m2 for patients with creatinine levels above institutional normal
  * Total serum bilirubin within normal institutional limits
  * ALT (SGPT) ≤ 2.5× the institutional upper limit of normal OR AST (SGOT) ≤ 2.5× the institutional upper limit of normal
* Ability to take medication sublingually
* Willingness and ability to comply with scheduled visits, laboratory tests, and other trial procedures
* Accessible for treatment and follow-up
* Female subjects: Use of two approved forms of contraceptives
* Male subjects: Use of two approved forms of contraceptives and willing to instruct their partners to use one form of contraceptive as well
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* MGMT promoter methylation status is positive (i.e., promoter is methylated)
* Prior radiotherapy for GBM within two (2) weeks of entering the study or has not recovered from adverse events due to agents administered more than four (4) weeks earlier
* Prior chemotherapy, immunotherapy, or radiation therapy for other cancers (except for treatment of limited curable skin cancers)
* Currently or recently (in the previous six months) part of a clinical trial involving any other investigational agents
* Hypersensitivity or allergy to any ingredient in the study drug
* Receiving any medications or substances that are known substantial inhibitors or inducers of CYP3A4
* Consumption of grapefruit or grapefruit juice three (3) days prior to screening or unwillingness to abstain from consuming grapefruit in any form during the study
* Uncontrolled intercurrent illness that would limit compliance with study requirements
* Pregnancy, possible pregnancy, plans for pregnancy, or active lactation or nursing
* Positive HIV or hepatitis status
* Unwillingness or inability to take medication sublingually
* Diagnosis of cancer more than 120 days prior to initial visit
* History of prior malignancy except curatively treated skin cancers
* History of prior chemotherapy or radiation for other cancers (except for treatment of limited curable skin cancers) before initial visit
* Clinically significant unstable medical conditions other than GBM
* Clinically relevant symptoms or clinically significant illness in the four (4) weeks prior to screening or registration, other than GBM
* Clinically significant unstable medical conditions, other than GBM, deemed by the investigator to pose an unacceptable risk to the patient
* History of substance abuse within the last two years
* Current use of recreational or medicinal cannabis, synthetic cannabinoid-based medications, or alcohol, or planned use while in the study
* Evidence of any diseases or conditions that may interfere with the study or interpretation of study results
* Inability or unwillingness to cooperate with the study procedures
* Known history of severe depression or psychiatric disorders, or active suicidal ideation
* Subjects with close affiliation with an investigational site
* Absence of or unwillingness to sign and date the informed consent document

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Through study completion, an average of one year
  The primary objective of this study is to evaluate the safety and tolerability of BRCX014 using clinical assessments and lab results.

SECONDARY OUTCOMES:
Maximum tolerated dose | Through study completion, an average of one year
  A secondary objective of this study is to identify the maximum tolerated dose of BRCX014.
Levels of metabolites | Through study completion, an average of one year
  A secondary objective of this study is to perform pharmacokinetics analyses by measuring the plasma concentrations of BRCX014, temozolomide, and their major metabolites using lab results.
Progression-free survival | Through study completion, an average of one year
  A secondary objective of this study is to measure PFS using lab results and radiographic data.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Avgeropoulos, MD, Principal Investigator — Orlando Health / UF Health Cancer Center

IPD SHARING:
Plan to Share IPD: No